CLINICAL TRIAL: NCT00629642
Title: A Randomized, Double Blind, Double Dummy, Placebo Controlled Study to Evaluate the Efficacy and Safety of Solifenacin Succinate (5 and 10mg Once Daily) Against Placebo and Oxybutynin Hydrochloride (5 mg Three Times Daily) in the Treatment of Subjects With Neurogenic Detrusor Overactivity
Brief Title: Clinical Study of Solifenacin Succinate in Patients With Bladder Symptoms Due to Spinal Cord Injury or Multiple Sclerosis
Acronym: SONIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 905-EC-005; 2006-005523-42 (Other: EudraCT)
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis; Neurogenic Bladder; Spinal Cord Diseases
Keywords: Neurogenic bladder; Vesicare
MeSH Terms: conditions — Multiple Sclerosis; Urinary Bladder, Neurogenic; Spinal Cord Diseases | interventions — Solifenacin Succinate; oxybutynin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- I.Solifenacin succinate 10mg (2x5mg 1/day) (Experimental): Oral
  Interventions: Drug: Solifenacin Succinate
- II.Solifenacin succinate 5mg (5mg 1/day) (Experimental): Oral
  Interventions: Drug: Solifenacin Succinate
- III.Oxybutynin hydrochloride 15mg (5mg 3/day) (Active Comparator): Oral
  Interventions: Drug: Oxybutynin Hydrochloride
- IV. Placebo (Placebo Comparator): Oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solifenacin Succinate — Oral, 10mg
  Other Names: Vesicare; YM905
  Arms: I.Solifenacin succinate 10mg (2x5mg 1/day)
Drug: Solifenacin Succinate — Oral, 5mg
  Other Names: Vesicare; YM905
  Arms: II.Solifenacin succinate 5mg (5mg 1/day)
Drug: Oxybutynin Hydrochloride — Oral, 15mg
  Arms: III.Oxybutynin hydrochloride 15mg (5mg 3/day)
Drug: Placebo — Oral
  Arms: IV. Placebo

SUMMARY:
A clinical study to evaluate the efficacy and safety of solifenacin in patients with bladder symptoms due to spinal cord injury or multiple sclerosis

DETAILED DESCRIPTION:
A clinical study to compare the efficacy and safety of solifenacin succinate in patients with neurogenic detrusor overactivity. In this randomized, double blind, double dummy study solifenacin will be compared to placebo and an active comparator, oxybutynin hydrochloride. Patients will be randomized to one of four treatment arms; solifenacin 10mg, solifenacin 5mg, placebo or oxybutynin 15mg. Patients will be assessed over a four week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been obtained
* Subjects with neurogenic detrusor overactivity due to:

  * Multiple sclerosis(MS)(EDSS≤8) or
  * Spinal cord injury(SCI)(partial or complete lesions)
* MS or SCI symptoms should be stable for >= 6 months
* Neurogenic detrusor overactivity symptoms should be stable for >= 6 months
* Subject is willing and able to perform clean, intermittent, catheterization, if required
* Subject is willing and able to take study medication in compliance with the protocol

Exclusion Criteria:

* Subjects with neurogenic detrusor overactivity due to Parkinson's or cerebrovascular disease
* Subjects with Sjögren's Syndrome or any similar symptoms
* Subjects with evidence of a symptomatic urinary tract infection, chronic inflammation such as interstitial cystitis, bladder stones, previous pelvic radiation therapy or previous or current malignant disease of the pelvic organs
* Subjects with stress incontinence or mixed incontinence where stress is the predominant factor as determined by the investigator
* Subjects with evidence of pressure sores >= grade 2
* Subjects with a history of bladder sphincterotomy
* Subjects with known history of vesico-ureteral reflux without upper urinary tract infection
* Any clinically significant condition, which in the opinion of the investigator makes the subject unsuitable for the study or includes a history of acute urinary retention, severe gastrointestinal obstruction (including paralytic ileus or intestinal atony), severe gastrointestinal conditions (including toxic megacolon or ulcerative colitis), myasthenia gravis, narrow angle glaucoma or shallow anterior chamber
* Subjects undergoing hemodialysis
* Subjects with severe hepatic impairment
* Concurrent use of drugs intended to treat symptoms of overactive bladder
* Use of antidepressants or muscle relaxants which have not been administered at a constant dose for >= 3 months
* Use of non-drug treatment intended to treat overactive bladder symptoms including electrostimulation therapy, botulinum toxin and vanilloids therapy in the six months prior to the commencement of the study
* Use of permanent, indwelling catheters
* Known or suspected hypersensitivity to solifenacin succinate, oxybutynin hydrochloride, other anti cholinergics or lactose
* Concomitant use of a strong CYP3A4 inhibitor, e.g. ketoconazole
* Pregnant women, women who intend to become pregnant during the study, women of childbearing potential who are sexually active and practicing an unreliable method of birth control or women who will be lactating during the study. Reliable contraceptive methods are intra-uterine devices, contraceptive pills of combination type, hormonal implants and injectable contraceptives
* Participation in any clinical study within 30 days of randomization, or the limit set by national law, whichever is longer
* Employees of the Astellas Group, third parties associated with the study, or the study site
* Subjects with maximum bladder capacity >= 400ml at visit 2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2008-03-14 (Actual); Primary Completion 2011-01-28 (Actual); Study Completion 2011-01-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in maximum cystometric capacity | 4 Weeks

SECONDARY OUTCOMES:
Change from baseline in bladder volume at first involuntary contraction | 4 Weeks
Change from baseline in pressure at first leak | 4 Weeks
Change from baseline in volume at first leak | 4 Weeks
Change from baseline in maximum detrusor pressure | 4 Weeks
Change from baseline in micturition or catheterization frequency | 4 Weeks
Change from baseline in incontinence episodes | 4 Weeks
Incidence and severity of adverse events | 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Department of (Neuro) Urology, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (38):
- Australia (4):
  - Brisbane
  - Melbourne
  - Perth
  - Randwick
- Belgium (6):
  - Antwerp
  - Esneux
  - Fraiture-en-Condroz
  - Ghent
  - Leuven
  - Melsbroek
- Czechia (3):
  - Brno
  - České Budějovice
  - Prague
- France (4):
  - Caen
  - Garches
  - Paris
  - Ploemeur
- Germany (4):
  - Berlin
  - Hagenow
  - Heidelberg
  - Kiel
- Hungary (3):
  - Nyíregyháza
  - Sopron
  - Szeged
- Italy (4):
  - Florence
  - Milan
  - Rome
  - Torino
- Netherlands (3):
  - Apeldoorn
  - Eindhoven
  - Nijmegen
- Saint Petersburg, Russia
- Spain (4):
  - Sant Joan d'Alacant, Alicante
  - Badalona, Barcelona
  - Getafe, Madrid
  - A Coruña
- United Kingdom (2):
  - Cardiff
  - Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- See also: Link to results on the Astellas Clinical Study Results website. — https://www.astellasclinicalstudyresults.com/study.aspx?ID=213